CLINICAL TRIAL: NCT00006503
Title: Prevalence & Progression of Subclinical Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 944; R01HL065581 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Coronary Arteriosclerosis; Carotid Artery Diseases; Menopause
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease; Carotid Artery Diseases

SUMMARY:
To evaluate subclinical atherosclerotic disease in menopausal women.

DETAILED DESCRIPTION:
BACKGROUND:

Decreased ovarian function and premenopausal obesity are likely the primary determinants of early coronary atherosclerosis as measured by calcification on EBCT. Aortic calcification occurs earlier than coronary calcification, may predict coronary calcification, and is expected to be the best marker of risk associated with traditional factors in these younger women. Preliminary data indicate that changes in coronary and aortic calcification can be observed over short periods of time in these women. A period of diminishing estrogen levels is the optimum time to observe changes in endothelial function which likely precede measurable atherosclerosis and thus may be the earliest markers for disease potential. Vascular stiffness, a marker for the biologic aging of the vascular system, is highly correlated with measures of insulin sensitivity which is altered in women at mid-life in conjunction with increases in central adiposity. Racial differences in disease prevalence and the relative importance of certain risk factors are likely.

DESIGN NARRATIVE:

Subclinical atherosclerosis will be evaluated in 728 women (305 African American, 423 Caucasian) enrolled in the Pittsburgh and Chicago sites of the Study of Women's Health Across the Nation (SWAN), a multicenter study characterizing the biological and psychosocial antecedents and sequellae of menopause. The extent to which diminishing ovarian function affects vascular function and accelerates the development of atherosclerosis in the coronary arteries, aorta and carotid arteries will be evaluated. Serial measures of coronary and aortic calcification (by electron beam computed tomography [EBCT] ), carotid atherosclerosis, endothelial function and aortic stiffening will be performed two years apart. The prevalence and progression of subclinical atherosclerosis will be evaluated in relation to serial measures of ovarian function, psychosocial and behavioral factors, markers of clotting and inflammation as well as traditional cardiovascular risk factors, all collected in SWAN. The study is conducted jointly by Dr. Lynda Powell (R01HL65581) at Rush-Presbyterian-St. Luke's Medical Center in Chicago and Dr. Kim Tyrrell (R01HL65591) at the University of Pittsburgh.

ELIGIBILITY:
No eligibility criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Powell — Rush-Presbyterian-St. Lukes Medical Center; Kim Tyrrell — University of Pittsburgh